CLINICAL TRIAL: NCT01875250
Title: A Phase II Trial of Enzalutamide in Combination With PSA-TRICOM in Patients With Non-Metastatic Castration Sensitive Prostate Cancer
Brief Title: Enzalutamide in Combination With PSA-TRICOM in Patients With Non-Metastatic Castration Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130153; 13-C-0153
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: Gene Transfer; Androgen Receptor Antagonist; PSA; Immune Response; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; rV-Tricom; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Enzalutamide for 3 months (Experimental): Enzalutamide for 3 months
  Interventions: Drug: Enzalutamide (Xtandi)
- Arm B - Enzalutamide for 3 months + PSA-TRICOM (Experimental): Enzalutamide 3 months + PSA-TRICOM (Prostvac-V/F) on weeks 1, 3, 5, 9,13,17 and 21
  Interventions: Biological: PROSTVAC-F (Fowlpox)/TRICOM; Biological: PROSTVAC-V (Vaccinia)/TRICOM; Drug: Enzalutamide (Xtandi)

INTERVENTIONS:
Biological: PROSTVAC-F (Fowlpox)/TRICOM — A recombinant fowlpox virus vector vaccine containing the genes for human prostate specific antigen (PSA) and three co-stimulatory molecules.
  Other Names: PROSTVAC-F/TRICOM
  Arms: Arm B - Enzalutamide for 3 months + PSA-TRICOM
Biological: PROSTVAC-V (Vaccinia)/TRICOM — A recombinant vaccinia virus vector vaccine containing the genes for human prostate specific antigen (PSA) and three co-stimulatory molecules.
  Other Names: PROSTVAC-V/TRICOM
  Arms: Arm B - Enzalutamide for 3 months + PSA-TRICOM
Drug: Enzalutamide (Xtandi) — An androgen receptor inhibitor.
  Other Names: Xtandi

SUMMARY:
Background:

- Enzalutamide is a well tolerated hormone therapy that is used to treat advanced prostate cancer. It is given to help kill cancer cells and limit cancer cell growth. A new possible way of treating prostate cancer is using a therapeutic cancer vaccine (immune stimulating therapy) that may help activate the immune system against the cancer. The immune stimulating vaccine will help white blood cells recognize and kill the cancer cells throughout the body. This vaccine therapy has been tested in hundreds of patients and is very well tolerated. Researchers want to see whether this vaccine, given with enzalutamide, is more effective at treating advanced prostate cancer than enzalutamide alone.

Objectives:

- To compare the safety and effectiveness of enzalutamide with and without vaccine therapy for advanced prostate cancer.

Key Eligibility:

* Men at least 18 years of age who have advanced castration sensitive prostate cancer.
* Patients must have testosterone within the normal range
* No evidence of metastatic prostate cancer on computed tomography (CT) or Bone scan
* No history of autoimmune diseases
* No previous immunotherapy within 3 years

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will be used to monitor the cancer before treatment.
* Participants will be separated into two groups. One group will have enzalutamide and the study vaccine. The other group will have enzalutamide alone.
* All participants will take enzalutamide once a day. They will take the drug for 3 months. This form of intermittent therapy is common in this population of patients.
* The vaccine group of participants will receive the new study vaccine. They will have a single injection on the first day of the first study cycle. There will be regular booster injections afterward. There will be one injection during the third week of treatment, and one in the fifth week. The vaccine will then be given every 4 weeks until 21 weeks have passed.
* Treatment will be monitored with frequent blood tests and imaging studies.

DETAILED DESCRIPTION:
Background:

* Androgen deprivation therapy (ADT) and surveillance are standard therapy options for prostate cancer patients with biochemical progression after localized therapy (or nonmetastatic castration sensitive prostate cancer; nmCSPC also known as D0 Prostate Cancer). These patients cannot be cured of prostate cancer and the primary therapeutic goal is to contain the disease with anti-androgen therapy.
* ADT can be administered intermittently consisting of multiple short courses or continuously with similar long-term clinical outcomes.
* Previous studies with high dose bicalutamide (androgen receptor antagonist, ARA) have shown significant biochemical control in nmCSPC.
* Enzalutamide is a modern ARA with greater androgen receptor affinity than bicalutamide and further impairs downstream effects of androgen receptor activation. This agent is FDA approved for the treatment of chemotherapy refractory metastatic castration resistant prostate cancer.
* Given its favorable side effect profile, there is strong interest in using enzalutamide to treat patients with earlier stages of prostate cancer including nmCSPC.
* PSA-TRICOM (Prostvac; developed by the National Cancer Institute [NCI] and licensed to Bavarian Nordic, Mountain View, California (CA)) is a novel candidate prostate cancer immunotherapy for the treatment of prostate cancer. It is a viral vector based therapeutic cancer vaccine that is administered via subcutaneous injections. In a randomized controlled Phase 2 trial, PSA-TRICOM therapy was associated with a prolongation of survival in men with metastatic castrate-resistant prostate cancer. A phase III trial is currently enrolling patients in this same population.
* There is also rationale to use therapeutic cancer vaccines such as PSA-TRICOM in earlier stage prostate cancer patients to maximize the potential therapeutic effect of immune stimulating therapy.
* An ongoing NCI clinical trial that combined PSA-TRICOM with flutamide (an older Food and Drug Administration (FDA) approved ARA) in nonmetastatic castration resistant prostate cancer has demonstrated safety and suggested the potential to improve time to progression.
* Analysis of previous trials using therapeutic cancer vaccines alone and in combination suggests that such therapies may alter tumor growth rate. If this hypothesis is correct, a therapeutic cancer vaccine may alter tumor regrowth rate/recovery after a cytoreductive therapy such as enzalutamide is discontinued.
* If PSA-TRICOM with enzalutamide can result in a reduced tumor regrowth rate as measured by PSA after a short course of enzalutamide therapy, it would provide an important proof of concept and potentially define it more clear role for therapeutic cancer vaccines in prostate cancer and potentially other cancers.
* To prospectively evaluate this hypothesis, all patients will be treated with enzalutamide in a manner similar to how short course ADT is used in common clinical practice. Half the patients will also be given PSA-TRICOM and PSA recovery after enzalutamide therapy will be compared between patients who received vaccine and those who did not.
* Preliminary data from the first cohort of randomized patients suggests that enzalutamide alone can induce an immunologic response. A second cohort of 15 patients will explore a lower dose of enzalutamide at 80 mg to determine if similar immunologic responses can also be seen at a lower dose, where toxicity is less likely.

Objectives:

Primary Endpoint:

-Determine if PSA-TRICOM combined with the novel androgen receptor antagonist enzalutamide will result in a decrease in PSA growth kinetics (tumor re-growth rate) after enzalutamide discontinuation in patients with non-metastatic, castration sensitive prostate cancer (i.e. patients with normal testosterone).

Eligibility:

* Patients with nonmetastatic castration sensitive prostate cancer and a PSA over 2.0 ng/ml
* Patients with normal testosterone levels.
* Histologically confirmed adenocarcinoma.
* Patients with a PSA doubling time of 12 months or less.
* Eastern Cooperative Oncology Group (ECOG) 0-1.

Design:

* Randomized pilot study
* Cohort 1:
* Thirty-four patients to be enrolled and randomized 1:1 to

  * Arm A: Enzalutamide for 3 months.
  * Arm B: Enzalutamide 3 months + PSA-TRICOM on weeks 1, 3,5,9,13,17 and 21.

Cohort 1:

* Arm A: Enzalutamide (n=17)
* Arm B: Enzalutamide + PSA-TRICOM (n=17)

  * Enzalutamide will be given at the standard dose of 160 mg daily for 3 months. PSATRICOM (Prostvac-V/F) will consist of a single subcutaneous (sc) immunization of Prostvac-V in Week 1, followed by 6 Prostvac-F immunizations administered in Weeks 3, 5, 9, 13, 17, and 21. Patients will be retreated with a 3-month course of enzalutamide after PSA has returned to baseline values at study entry or higher. Patients will have had to be on study for at least 7 months or longer in order to be retreated with an additional course of enzalutamide therapy. Patients will be followed for PSA recovery after enzalutamide has been discontinued. Patients who do not develop a 25% decline in PSA after 3 months will not be evaluated for tumor re-growth and additional patients will be enrolled to evaluate for that endpoint. Patients will be stratified based on a doubling time of greater than or less than 6 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histopathological documentation of prostate cancer confirmed in the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center, or Walter Reed National Military Medical Center prior to enrollment. If no pathologic specimen is available, patients may enroll with a pathologists report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.

B. Biochemical progression defined as follows:

* For patients following definitive radiation therapy: a rise in prostate-specific antigen (PSA) of greater than or equal to 2 ng/mL above the nadir (per Radiation Therapy Oncology Group (RTOG)-American Society for Therapeutic Radiology and Oncology (ASTRO) consensus criteria).
* For patients following radical prostatectomy: rising PSA after surgical procedure. (Patients must have a PSA greater than or equal to 2ng/ml)

C. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky greater than or equal to 80%).

D. Patients must have a PSA doubling time of 12 months or less.

E. Patients must have a rising PSA as confirmed by 3 values done at least 1 week apart and over no less than 1 month.

F. Recovery from acute toxicity related to prior therapy, including surgery and radiation, or no toxicity greater than or equal to grade 2.

G. Negative computed tomography (CT) scan/magnetic resonance imaging (MRI) and bone scan for metastatic prostate cancer.

H. Hematological eligibility parameters (within 16 days before starting therapy):

Granulocyte count greater than or equal to 1000/mm(3)

Platelet count greater than or equal to 100,000/mm(3)

Hemoglobin (Hgb) greater than or equal to 10 g/dL

I. Biochemical eligibility parameters (within 16 days before starting therapy):

Hepatic function: bilirubin less than or equal to 1.5 mg/dL (OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0), aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 2.5 times upper limit of normal.

J. No other active malignancies within the past 36 months (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder) or life-threatening illnesses

K. Willing to travel to the National Institutes of Health (NIH) for follow-up visits.

L. 18 years of age or older.

M. Able to understand and sign informed consent.

N. Baseline testosterone greater than or equal to lower limit of normal.

O. PSA less than or equal to 20 ng/mL.

P. The effects of enzalutamide, PSA-TRICOM or the combination on the developing human fetus are unknown. For this reason, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

A. Immunocompromised status due to:

* Human immunodeficiency virus (HIV) positivity.
* Active autoimmune diseases such as Addison's disease, Hashimoto s thyroiditis, systemic lupus erythematosus, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Graves disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including central nervous system (CNS), heart, lungs, kidneys, skin, and gastrointestinal (GI) tract will be allowed.
* Other immunodeficiency diseases

B. Chronic administration (defined as daily or every other day for continued use greater than 14 days) of corticosteroids deemed systemic by investigator within 28 days before the first planned dose of PSA-TRICOM. Use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed.

C. Serious intercurrent medical illness that, in the judgment of the investigator, would interfere with patient's ability to carry out the treatment program.

D. History of seizure, including any febrile seizure, loss of consciousness, or transient ischemic attack, or any condition that may pre-dispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization).

E. Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (eg phytoestrogens and saw palmetto)

F. History of prior chemotherapy

G. History of prior immunotherapy within the last 3 years

H. Major surgery within 4 weeks prior to enrollment (Day 1 visit).

I. History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide or poxviral vaccines (e.g., vaccinia vaccine)

J. Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin).

K. History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis

L. Previous serious adverse reactions to smallpox vaccination

M. Unable to avoid close contact or household contact with the following highrisk individuals for three weeks after the Day 1 vaccination: (a) children 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczematoid skin disorders, or (d) immunocompromised individuals, such as those with human immunodeficiency virus (HIV).

N. Receipt of an investigational agent within 30 days (or 60 days for an antibody based therapy) before the first planned dose of study drugs.

O. Patients who test positive for Hepatitis B virus (HBV) or hepatitis C virus (HCV)

P. Use of herbal products that may decrease PSA levels (e.g. saw palmetto)

Q. Any gastrointestinal disease that could hinder the absorption of enzalutamide

R. Uncontrolled hypertension (Systolic Blood Pressure (SBP)>170/ Diastolic Blood Pressure (DBP)>105)

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furr BJ. "Casodex" (ICI 176,334)--a new, pure, peripherally-selective anti-androgen: preclinical studies. Horm Res. 1989;32 Suppl 1:69-76. doi: 10.1159/000181315. PMID 2533159
- [Background] Chen Y, Clegg NJ, Scher HI. Anti-androgens and androgen-depleting therapies in prostate cancer: new agents for an established target. Lancet Oncol. 2009 Oct;10(10):981-91. doi: 10.1016/S1470-2045(09)70229-3. PMID 19796750
- [Background] Sartor AO, Tangen CM, Hussain MH, Eisenberger MA, Parab M, Fontana JA, Chapman RA, Mills GM, Raghavan D, Crawford ED; Southwest Oncology Group. Antiandrogen withdrawal in castrate-refractory prostate cancer: a Southwest Oncology Group trial (SWOG 9426). Cancer. 2008 Jun;112(11):2393-400. doi: 10.1002/cncr.23473. PMID 18383517
- [Derived] Madan RA, Karzai F, Donahue RN, Al-Harthy M, Bilusic M, Rosner II, Singh H, Arlen PM, Theoret MR, Marte JL, Cordes L, Couvillon A, Hankin A, Williams M, Owens H, Lochrin SE, Chau CH, Steinberg S, Figg WD, Dahut W, Schlom J, Gulley JL. Clinical and immunologic impact of short-course enzalutamide alone and with immunotherapy in non-metastatic castration sensitive prostate cancer. J Immunother Cancer. 2021 Mar;9(3):e001556. doi: 10.1136/jitc-2020-001556. PMID 33664086
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0153.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM
Started | 19 | 19
Completed | 17 | 19
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 20
  >=65 years | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.46) | 66.07 (5.29) | 65.88 (6.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Tumor Growth Rate
Description: Growth rate was measured using the growth rate equation -f(t) = exp (-d*t) + exp (g*t) -1 where exp is the base of the natural algorithm, e = 2.7182 and t is days since treatment started. The tumor growth rate equation measures Prostate Specific Antigen (PSA) rise over time. The UOM is unitless because this is a way to measure PSA kinetics.
Time Frame: 7 months
Measure: Number; unit: unitless
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM
Number analyzed (Participants) | 19 | 19
unitless | 0.031 | 0.030
Statistical Analysis 1: Comparison: Arm A - Enzalutamide for 3 Months vs Arm B - Enzalutamide for 3 Months + PSA-TRICOM; Test type: Superiority; p = 0.74, Wilcoxon rank sum tests

2. Secondary Outcome: Mean Pretreatment Plasma Vascular Endothelial Growth Factor (VEGF) Concentration 30 Days After the Start of Course 1 and Course 2 of Enzalutamide
Description: VEGF was measured by the enzyme-linked immunosorbent assay (ELISA) assay. The lower limit of quantitation of assay was 9.0 pg/ml.
Time Frame: 30 Days After the Start of Course 1 and Course 2 of Enzalutamide
Population: It was pre-specified to combine analysis for Arms of growth factors.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- All Participants: All participants who received Enzalutamide for 3 months and Enzalutamide 3 months + PSA-TRICOM.
Arm/Group | All Participants
Number analyzed (Participants) | 36
pg/ml
  Course 1 | 192 (82)
  Course 2 | 165.04 (82.38)

3. Secondary Outcome: Median Testosterone After 84 Days of Enzalutamide
Description: Normal testosterone is 270-1070 nd/dL.
Time Frame: 84 days
Population: It was pre-specified to combine analysis for testosterone. In addition, data was not analyzed beyond Course 1 because it was not part of the initial statistical plan.
Measure: Median (Full Range); unit: ng/dl
Groups:
- All Participants: All participants who received Enzalutamide for 3 months and Enzalutamide 3 months + PSA-TRICOM,
Arm/Group | All Participants
Number analyzed (Participants) | 36
ng/dl | 834 [308 to 1579]

4. Secondary Outcome: Percent Change in Prostate Specific Antigen (PSA) After 84 Days of Enzalutamide in Course 1
Description: Median PSA change would be considered optimal.
Time Frame: 84 days
Measure: Median (Full Range); unit: Percent change
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM
Number analyzed (Participants) | 19 | 19
Percent change | -99 [-84 to -99] | -99 [-87 to -99]

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 43 months and 13 days for Arm A, and 78 months and 6 days for Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM
Number analyzed (Participants) | 19 | 19
Participants | 19 | 19

6. Secondary Outcome: Median Time Until Prostate Specific Antigen (PSA) Recovery From Baseline Following Course 1 and Course 2 of Enzalutamide
Description: PSA recovery is defined as the return above baseline PSA in participants with normal testosterone and non-metastatic, castration sensitive prostate cancer.
Time Frame: up to 41 months
Population: It was pre-specified to combine analysis for Arms of PSA Recovery time.
Measure: Median (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 36
Days
  Course 1 | 224 [84 to 1246]
  Course 2 | 189 [78 to 400]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 43 months and 13 days for Arm A, and 78 months and 6 days for Arm B.
Arm/Group | Arm A - Enzalutamide for 3 Months | Arm B - Enzalutamide for 3 Months + PSA-TRICOM
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Enzalutamide for 3 Months (N=19) | Arm B - Enzalutamide for 3 Months + PSA-TRICOM (N=19)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Surgical biopsy 1/5 and 6 weeks of radiation scheduled to start January 2017.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Enzalutamide for 3 Months (N=19) | Arm B - Enzalutamide for 3 Months + PSA-TRICOM (N=19)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (9) | 5 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (6) | 8 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 2 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (12)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Breast atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 15 (19) | 16 (21)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 4 (10) | 4 (5)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (2) | 3 (7)
Cholesterol high (Investigations) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Creatinine increased (Investigations) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (10) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 5 (6) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Diplopia Lightheadedness intermittent (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Tearfullness (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (26) | 16 (28)
Fever (General disorders) | 0 (0) | 1 (3)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Flatulence (General disorders) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 6 (7)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal disorders - Other, Damaged broken tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 9 (13) | 7 (8)
Headache (Nervous system disorders) | 2 (2) | 6 (13)
Hematuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 3 (4) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (26) | 8 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 4 (6) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (26) | 7 (24)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Infections and infestations - Diverticulitis-received 2 antibiotics (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Flu 2-3 weeks ago, (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, No antibiotics (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, URI and rash (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, URI-head cold, uses Dayquil (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, UTI (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Cold (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Cold- OTC meds (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Erythema (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, Fungal infection-Terbinafine (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, URI- no antibiotics (Infections and infestations) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 18 (70)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (2) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 3 (4) | 4 (4)
Libido decreased (Reproductive system and breast disorders) | 1 (1) | 3 (4)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (15) | 8 (22)
Memory impairment (Nervous system disorders) | 1 (1) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 2 (4)
Nipple deformity (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 4 (6) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 4 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Fullness B/L in temporal area-not painful (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Pre cancerous lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Sores on feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Abraasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Allergic reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Callus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cold sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3)
Weight gain (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 5 (9) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT01875250/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT01875250/ICF_001.pdf